CLINICAL TRIAL: NCT01541865
Title: Treatment of Resistant Hypertension Using a Radiofrequency Percutaneous Transluminal Angioplasty Catheter (REDUCE-HTN) - POST MARKET APPROVAL CLINICAL SURVEILLANCE STUDY
Brief Title: Treatment of Resistant Hypertension Using a Radiofrequency Percutaneous Transluminal Angioplasty Catheter
Acronym: REDUCE-HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002-020
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: hypertension, renal denervation, uncontrolled hypertension, medication resistant hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Denvervation (Other): All subjects who meet the inclusion criteria and are enrolled in this trial will be treated with the Vessix Renal Denervation System.
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation — percutaneous renal denervation using the Vessix RF balloon catheter
  Other Names: Vessix V2 Renal Denervation System

SUMMARY:
The Study objective is to assess the performance of the Vessix V2 Renal Denervation System for the treatment of uncontrolled hypertension using an innovative percutaneous Radio Frequency (RF) balloon catheter renal denervation device.

DETAILED DESCRIPTION:
This study will evaluate the hypothesis that the Vessix V2 Renal Denervation System can be employed to reduce systolic and diastolic blood pressure at 6 months as compared to pre-treatment baseline blood pressures.

Patient blood pressure will be measured by in the office according to recognized international techniques and standards.

Procedural success shall be defined as ability to complete the renal denervation treatment using the V2 balloon catheter device and RF generator.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have provided written informed consent;
2. Subjects who are ≥ 18 years and ≤ 75 years of age;
3. Subjects who have Systolic Blood Pressure (SBP) ≥ 160 mm Hg based on an average of three (3) office-based blood pressure readings (seated) measured according to protocol;
4. Subjects with ≥ 3 anti-hypertensive drugs at maximally tolerated doses with stable regimen for at least 2 weeks prior to enrollment
5. Subjects with a estimated glomerular filtration rate (eGFR) ≥ 45 ml/min/1.73m^2;
6. Suitable renal artery anatomy
7. Subjects who are willing and able to comply with all study procedures.

Exclusion Criteria:

1. Subjects with known/diagnosed secondary hypertension;
2. Subjects who are contraindicated for anticoagulation medications (heparin, aspirin, Angiomax, etc.), analgesic medications (morphine, fentanyl, etc.), anxiolytic medications (alprazolam, lorazepam, diazepam, etc.) or other medications required for an interventional procedure;
3. Subjects with known bleeding or hyper-coagulation disorders;
4. Subjects who have type 1 diabetes mellitus;
5. Subjects who have experienced a myocardial infarction, unstable angina pectoris, uncompensated heart failure, or a cerebrovascular accident within six (6) months prior to the screening visit, or have widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques;
6. Subjects who have planned percutaneous vascular or surgical intervention for any reason within the next 6 months;
7. Subjects who have hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous;
8. Subjects who have an implantable cardioverter defibrillator, pacemaker, or clinically significant abnormal electrocardiogram
9. Subjects who have any serious medical condition, which in the opinion of the investigator, may adversely affect patient safety or the efficacy of the procedure in the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, or significant anemia);
10. Subjects who are pregnant, nursing or planning to become pregnant;
11. Subjects who have a known, unresolved history of drug use or alcohol abuse/dependency;
12. Subjects who are currently enrolled in any investigational study wherein patient participation has not been completed;
13. Subjects who, for any reason, may not be able to understand or comply with instructions;
14. Subjects who are contraindicated for intravascular contrast material;
15. Subjects who are currently taking estrogen or any estrogen-like compound.
16. Subjects who have had a prior renal denervation procedure
17. Subjects with prior intervention to right or left renal artery;
18. Subjects with ≥ 30% renal artery stenosis
19. Subjects with severe femoral, renal, iliac or aortic calcification that may cause a potential complication at the time of the procedure;
20. Subjects in which the physician is unable to safely cannulate the renal artery;
21. Subjects in which the physician is unable to percutaneously access the femoral artery;
22. Subjects with one kidney.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, M.D., Principal Investigator — CardioVascular Center Frankfurt, Germany
Locations (26):
- Australia (5):
  - St. Vincent's Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Cardiology Clinical Research Centre, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Cardiovascular Research Centre (Monash Heart), Clayton, Victoria
- Austria (2):
  - AKH Linz, Linz
  - Salzburger Landeskliniken Universitats Krankenhaus, Salzburg
- Belgium (2):
  - OLV Ziekenhuis, Aalst
  - Cliniques Universiaires Saint-Luc, Brussels
- France (2):
  - Hôpital Européen Georges Pompidou, Paris
  - Clinic Pasteur, Toulouse
- Germany (9):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Kardiologische Praxis Main-Taunus, Bad Soden/Taunus
  - Vascular Center Berlin, Ev. Königin Elisabeth Hospital, Berlin
  - St. Vincenz Krankenhaus Abt. Kardiologie, Essen
  - CardioVascular Center, Sankt Katharinen Krakenhaus, Frankfurt
  - Hamburg University Cardiovascular Center, Hamburg
  - Saarland University Hospital Department of Internal Medicine III Non-surgical Intensive Care, Cardiology and Angiology, Homburg/Saar
  - University Leipzig, Leipzig
  - German Heart Center Munich, Münich
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Erasmus Medical Center-Thorax Center, Rotterdam
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Mercy Angiography Unit Ltd, Auckland
- Switzerland (2):
  - University Hospital of Geneva, Cardiology Center, Geneva
  - Switzerland University Hospital Clinic for Cardiology, Zurich

REFERENCES:
- [Result] Sievert H, Schofer J, Ormiston J, Hoppe UC, Meredith IT, Walters DL, Azizi M, Diaz-Cartelle J, Cohen-Mazor M. Renal denervation with a percutaneous bipolar radiofrequency balloon catheter in patients with resistant hypertension: 6-month results from the REDUCE-HTN clinical study. EuroIntervention. 2015 Feb;10(10):1213-20. doi: 10.4244/EIJY14M12_01. PMID 25452197
- [Result] Persu A, Sapoval M, Azizi M, Monge M, Danse E, Hammer F, Renkin J. Renal artery stenosis following renal denervation: a matter of concern. J Hypertens. 2014 Oct;32(10):2101-5. doi: 10.1097/HJH.0000000000000323. No abstract available. PMID 25186534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of up to 150 subjects was planned; 146 subjects were enrolled at 23 centers in the Europe, Australia and New Zealand from February 22, 2012 to April 8, 2013.
Groups:
- Renal Denervation: All subjects who meet the inclusion criteria and are enrolled in this trial will be treated with the Vessix Renal Denervation System.
Period: Overall Study
Arm/Group | Renal Denervation
Started | 146
Completed | 124
Not Completed | 22
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 89
Race/Ethnicity, Customized [Number; unit: participants]
  White | 135
  Black, Asian, Other | 11
Region of Enrollment [Number; unit: participants]
  New Zealand | 21
  Austria | 13
  Netherlands | 5
  Belgium | 17
  Australia | 31
  France | 8
  Switzerland | 2
  Germany | 49
Type 2 Diabetes [Number; unit: participants]
  Type 2 Diabetes | 41
  Non-Diabetic | 105
Coronary Artery Disease [Number; unit: participants]
  Coronary Artery Disease | 55
  No Coronary Artery Disease | 91
Congestive Heart Failure [Number; unit: participants]
  Congestive Heart Failure | 3
  No Congestive Heart Failure | 143
Dyslipidemia [Number; unit: participants]
  Dyslipidemia | 85
  No Dyslipidemia | 61
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 182.4 (18.4)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 100.2 (14.0)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 71.7 (14.8)
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 82.7 (22.5)
Serum Creatinine [Mean (Standard Deviation); unit: micromol/L] | 82.0 (20.0)
Number of Antihypertensive Medications per Patient [Mean (Standard Deviation); unit: Antihypertensive Medications per Patient] | 4.8 (1.5)
Antihypertensive Medications [Number; unit: participants]
  Subjects on greater than or equal to 5 medications | 79
  Subjects on 4 medications | 38
  Subjects on 3 medications | 26
  Subjects on 2 medications | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Blood Pressure at Six (6) Months as Measured by Office-based Blood Pressure Assessment
Description: Change in systolic and diastolic blood pressure at six (6) months as measured by office-based blood pressure assessment following therapeutic renal denervation compared to baseline. Office blood pressure will be measured using a validated electronic device according to a standardized procedure. .
Time Frame: Baseline and 6 months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 3 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 143
mm Hg
  Systolic | -24.5 (22.1)
  Diastolic | -10.3 (12.7)

2. Secondary Outcome: Absence of Flow Limiting Stenosis in the Renal Artery
Description: Absence of flow limiting stenosis in the renal artery at six (6) months follow up time point as measured by renal duplex ultrasound
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants w/o flow limiting stenosis
Arm/Group | Renal Denervation
Number analyzed (Participants) | 143
participants w/o flow limiting stenosis | 139

3. Primary Outcome: Change in Systolic and Diastolic Blood Pressure at Six (6) Months as Measured by 24-hour Ambulatory Blood Pressure
Description: Change in systolic and diastolic blood pressure at six (6) months as measured by 24-hour ambulatory blood pressure monitoring (ABPM) following therapeutic renal denervation compared to baseline using a validated ABPM device.
Time Frame: Baseline and 6 months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 76 participants were not evaluable at either the baseline or 6 month assessment.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 70
mm Hg
  Systolic | -8.0 (14.6)
  Diastolic | -5.7 (9.2)

4. Secondary Outcome: Renal Artery Dissection or Perforation During the Procedure That Requires Stenting or Surgery
Time Frame: Duration of the procedure (average of 65 minutes)
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
participants | 0

5. Secondary Outcome: Renal Artery Infarction or Embolus
Time Frame: Duration of the procedure (average of 65 minutes)
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
participants | 0

6. Secondary Outcome: Cerebrovascular Accident (CVA) at Time of Procedure
Time Frame: Duration of the procedure (average of 65 minutes)
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
participants | 0

7. Secondary Outcome: Myocardial Infarction at Time of Procedure
Time Frame: Duration of the procedure (average of 65 minutes)
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
participants | 0

8. Secondary Outcome: Sudden Cardiac Death at Time of Procedure
Time Frame: Duration of the procedure (average of 65 minutes)
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 146
participants | 0

9. Secondary Outcome: Angiographically-documented Renal Stenosis Requiring an Intervention
Time Frame: 2 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 22 participants were not evaluable.
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 124
participants | 1

10. Secondary Outcome: Chronic Symptomatic Orthostatic Hypotension
Time Frame: 2 Years
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 124
participants | 0

11. Secondary Outcome: Hypertensive Emergency Necessitating Hospital Admission (Unrelated to Medication and/or Non-compliance)
Time Frame: 2 Years
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 124
participants | 10

12. Secondary Outcome: Reduction in Estimated Glomerular Filtration Rate (eGFR) >25%
Time Frame: 2 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 25 participants were not evaluable.
Measure: Number; unit: participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 121
participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collect through the 2 year follow up visit.
Arm/Group | Renal Denervation
Serious Adverse Events (participants affected / at risk) | 69/146
Other Adverse Events (participants affected / at risk) | 70/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=146)
Access Site Infection (Surgical and medical procedures) | 2 (2) — Procedure Related
Clot or Thrombus Formation (Surgical and medical procedures) | 1 (1) — Procedure Related
Hematoma (Surgical and medical procedures) | 1 (1) — Procedure Related
Other Vascular - Stenosis (Surgical and medical procedures) | 1 (1) — Device Related/Procedure Related
Pseudoaneurysm (Surgical and medical procedures) | 1 (1) — Procedure Related
Other - Flank Pain (Surgical and medical procedures) | 1 (1) — Procedure Related
Other - Digestive (vomiting) (Surgical and medical procedures) | 1 (1) — Procedure Related
Other - Hypertensive Crisis (Surgical and medical procedures) | 4 (5) — Device Related/Procedure Related
Other Cardiac - Hypertensive episode (Surgical and medical procedures) | 1 (2) — Device Related
Acute Occlusion/Vessel Closure (Surgical and medical procedures) | 1 (1)
Stent Required (Surgical and medical procedures) | 1 (1)
Other Vascular - Carotid Stenosis (Vascular disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 4 (6)
Other Renal - Renal Calcification (Vascular disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other Pulmonary (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Other Infectious/Inflammatory (Infections and infestations) | 9 (10)
Stroke (Vascular disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 5 (8)
Other Neurological (General disorders) | 2 (2)
Unanticipated Adverse Events - Prolapsis Uteri (Reproductive system and breast disorders) | 1 (1)
Other Cardiac - Chest Pain/Angina (Cardiac disorders) | 7 (8)
Other - Hypertension (Renal and urinary disorders) | 13 (21)
Other Cardiac - Fibrillation (Cardiac disorders) | 5 (5)
Other Cardiac - Tachycardia (Cardiac disorders) | 1 (1)
Other - Inflammation/Infection (Infections and infestations) | 10 (14)
Other - Thoracic/Abdominal Pain (General disorders) | 4 (4)
Other - Hernia (General disorders) | 1 (1)
Other - Gastrointestinal/Rectal (Gastrointestinal disorders) | 6 (7)
Other - Skeletal/Connective Tissue (Musculoskeletal and connective tissue disorders) | 13 (19)
Other - Deconditioning post medical illness (General disorders) | 1 (1)
Other - Dementia (General disorders) | 1 (1)
Other - Diabetes (Metabolism and nutrition disorders) | 5 (6)
Other - Elective Surgery (Surgical and medical procedures) | 2 (2)
Other - Priapismus (Reproductive system and breast disorders) | 1 (1)
Other - Limb oedema/ Ulceration (Vascular disorders) | 2 (2)
Other - Coronary Sub-Occlusion (Vascular disorders) | 1 (1)
Other - Nausea (General disorders) | 1 (1)
Other - Overdose (General disorders) | 1 (1)
Other - Prostate Carcinoma (Reproductive system and breast disorders) | 1 (1)
Other - Sleep Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other - Suicide Ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=146)
Access Site Complications (Skin and subcutaneous tissue disorders) | 20 (22) — Procedure Related
Pain (General disorders) | 23 (23) — Procedure Related
Hematoma (Skin and subcutaneous tissue disorders) | 18 (19) — Procedure Related
Anaesthesia Related - Nausea/Vomiting (General disorders) | 12 (14) — Procedure Related
Reduced Kidney Function (Renal and urinary disorders) | 9 (9) — Device Related
Dizziness (General disorders) | 16 (18) — Potentially Related to Device and/or Procedure
Hypertension (General disorders) | 14 (14) — Potentially Related to Device and/or Procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No